CLINICAL TRIAL: NCT07288619
Title: Evaluation of the Clinical Effectiveness of Nutritional Supplements in Pulmonary Cachexia: A Quasi-Experimental Trial of n-3 PUFAs and Vitamin D
Brief Title: Therapeutic Efficacy of Nutritional Supplementation in Cachexia Associated With Chronic Pulmonary Disease
Acronym: CATCH-PulMo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Safeer Khan (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Sponsor-Investigator, Safeer Khan, Principal Investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAMC/IRB/EA112025
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Cachexia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cachexia | interventions — Fatty Acids, Omega-3; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- N-3 Polyunsaturated Fatty Acids (PUFA) (Experimental)
  Interventions: Dietary Supplement: N-3 Polyunsaturated Fatty Acids (PUFA)
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: N-3 Polyunsaturated Fatty Acids (PUFA) — Dosage, 1000 mg per dose; Frequency, Twice daily (BID); Duration, Six weeks; Administration Route, Oral softgel capsule; Manufacturer, Donated by NOW Foods (Bloomingdale, Illinois, USA).
  Arms: N-3 Polyunsaturated Fatty Acids (PUFA)
Dietary Supplement: Vitamin D — Dosage, 1000 IU per dose (total 2000 IU per day); Frequency, Twice daily (BID); Duration, Six weeks; Administration Route, Oral softgel capsule; Manufacturer, Donated by NOW Foods (Bloomingdale, Illinois, USA).
  Arms: Vitamin D

SUMMARY:
Pulmonary cachexia, observed in individuals with chronic obstructive pulmonary disease (COPD) is a multifactorial syndrome characterized by disruptions in energy metabolism, increased protein degradation, and an impaired capacity to preserve muscle mass. These metabolic disturbances not only exacerbate the underlying respiratory condition but also significantly contribute to elevated mortality rates among affected individuals.

Current therapeutic strategies for managing cachexia primarily emphasize pharmacological treatments, nutritional interventions, and multimodal approaches. Among the nutritional interventions, various supplements have shown potential in mitigating the catabolic processes associated with cachexia. Notably, supplementation with n-3 polyunsaturated fatty acids (n-3 PUFAs) and vitamin D has emerged as a promising intervention, likely due to their involvement in key pathological mechanisms underlying the disease.

While previous studies have investigated the combined effects of these supplements through oral nutritional supplementation, this study aims to evaluate and compare the clinical effectiveness of n-3 PUFAs and vitamin D as distinct therapeutic interventions for managing pulmonary cachexia.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide both written and verbal consent.
2. Clinically diagnosed with chronic obstructive pulmonary disease (COPD).
3. Diagnosis of pulmonary cachexia according to Cachexia Consensus Conference criteria

Exclusion Criteria:

1. Patients experiencing acute exacerbations of COPD.
2. Patients with co-morbid chronic diseases that can also cause cachexia, including cancer, HIV/AIDS, heart failure, chronic renal failure, liver cirrhosis, and rheumatoid arthritis
3. Pregnant women and patients with abnormal liver and/or renal function tests.
4. Patients who have taken n-3 PUFAs, Vitamin D, or any intervention for cachexia in the past four weeks.
5. Patients on oral or parenteral corticosteroids for more than four weeks.
6. Patients with a history of allergies to fish-derived products, n-3 polyunsaturated fatty acids (PUFAs), or Vitamin D.
7. Patients with a metabolic disorder that can lead to changes in body composition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and Week 6
  Change in BMI from baseline (pre-intervention), measured using a calibrated weight and height scale, and expressed in kg/m².
Fat-Free Mass Index (FFMI) | Baseline and week 6
  Change in FFMI from baseline (pre-intervention), measured using bioelectrical impedance analysis, and expressed in kg/m².
Fat Mass Index (FMI) | Baseline and week 6
  Change in FFM from baseline (pre-intervention), measured using bioelectrical impedance analysis, and expressed in kg/m².
Handgrip Strength (HGS) | Baseline and week 6
  Change from baseline HGS measured in kilograms using a calibrated dynamometer.
Mid-Arm Muscle Circumference (MAMC) | Baseline and week 6
  Change in MAMC from baseline (pre-intervention), calculated using the formula: MAMC = Mid-Arm Circumference (MAC) - (π × Triceps Skinfold (TSF)), expressed in centimeters (cm). The Mid-Arm Circumference (MAC) is measured using a flexible tape measure at the midpoint of the upper arm, and Triceps Skinfold (TSF) is measured using skinfold caliper.
Simplified Nutritional Appetite Questionnaire (SNAQ) - Anorexia | Baseline and week 6
  Change in SNAQ score from baseline (pre-intervention). SNAQ is a brief, four-item screening tool used to assess anorexia with a score of 14 or below indicates poor appetite.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Baseline and week 6
  Change in FACIT-F score from baseline (pre-intervention). FACIT-F is a 13-item scale used to assess the severity of fatigue in patients with chronic illnesses, with a scale range of 0 to 52. Higher scores indicate less fatigue (better functional status), while lower scores indicate more severe fatigue (worse functional status).
Edmonton Symptom Assessment System (ESAS) - Symptom Burden | Baseline and week 6
  Change in ESAS score from baseline (pre-intervention). ESAS is a multi-item scale used to assess symptom burden in patients. The scale ranges from 0 to 100, with higher scores indicating greater symptom severity and lower scores indicating less severe symptoms

SECONDARY OUTCOMES:
Medication Adherence | Week 6
  Percentage of patients achieving medication adherence of 80% or more, as assessed through pill count.
Adverse Effects | Eight weeks
  Percentage of patients experiencing adverse effects, assessed throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulab Devi Teaching Hospital, Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolodny GM. Patterns of protein synthesis in the HeLa cancer cell. Am J Roentgenol Radium Ther Nucl Med. 1969 Apr;105(4):746-55. doi: 10.2214/ajr.105.4.746. No abstract available. PMID 5803606
- [Background] van Beers M, Rutten-van Molken MPMH, van de Bool C, Boland M, Kremers SPJ, Franssen FME, van Helvoort A, Gosker HR, Wouters EF, Schols AMWJ. Clinical outcome and cost-effectiveness of a 1-year nutritional intervention programme in COPD patients with low muscle mass: The randomized controlled NUTRAIN trial. Clin Nutr. 2020 Feb;39(2):405-413. doi: 10.1016/j.clnu.2019.03.001. Epub 2019 Mar 18. PMID 30954363